CLINICAL TRIAL: NCT02661490
Title: A Phase II, Randomized, Double-blind, Safety and Immunogenicity Trial of Norovirus GI.1/GII.4 Bivalent Virus-Like Particle Vaccine in Healthy Elderly Adults
Brief Title: Safety and Immunogenicity of Norovirus GI.1/GII.4 Bivalent Virus-Like Particle Vaccine in an Elderly Population
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NOR-204; U1111-1162-4913 (Registry Identifier: WHO)
Record Dates: First submitted 2016-01-08; First posted 2016-01-22 (Estimated); Results first posted 2020-05-18 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-04

CONDITIONS: Norovirus
Keywords: Norovirus
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Arm 1: NoV Vaccine Formulation A _1-Dose (Experimental): Participants ≥ 60 years of age, 1-dose regimen: Norovirus bivalent placebo-matching vaccine, intramuscularly (IM), on Day 1, followed by norovirus (NoV) GI.1 (15 μg)/GII.4 (50 μg) bivalent virus-like particle (VLP) vaccine (Formulation A), IM, on Day 29.
  Interventions: Biological: Norovirus GI.1/GII.4 Bivalent VLP Vaccine; Drug: 0.9% sodium chloride (saline)
- Arm 2: NoV Vaccine Formulation A _2-Dose (Experimental): Participants ≥ 60 years of age, 2-dose regimen: Norovirus GI.1 (15 μg)/GII.4 (50 μg) bivalent VLP vaccine (Formulation A), IM, on Days 1 and 29.
  Interventions: Biological: Norovirus GI.1/GII.4 Bivalent VLP Vaccine
- Arm 3: NoV Vaccine Formulation B_1-Dose (Experimental): Participants ≥ 60 years of age, 1-dose regimen: Norovirus bivalent placebo-matching vaccine, IM on Day 1, followed by norovirus GI.1 (15 μg)/GII.4 (50 μg) bivalent VLP vaccine with 15 μg monophosphoryl lipid A (MPL) (Formulation B), IM, on Day 29.
  Interventions: Drug: 0.9% sodium chloride (saline); Biological: Norovirus GI.1/GII.4 Bivalent VLP Vaccine
- Arm 4: NoV Vaccine Formulation B_2-Dose (Experimental): Participants ≥ 60 years of age, 2-dose regimen: Norovirus GI.1 (15 μg)/GII.4 (50 μg) bivalent VLP vaccine with 15 μg MPL (Formulation B), IM, on Days 1 and 29.
  Interventions: Biological: Norovirus GI.1/GII.4 Bivalent VLP Vaccine
- Arm 5: NoV Vaccine Formulation A_1-Dose (Experimental): Participants 18 to 49 years of age, 1-dose regimen: Norovirus bivalent placebo-matching vaccine, IM, on Day 1, followed by norovirus GI.1 (15 μg)/GII.4 (50 μg) bivalent VLP vaccine (Formulation A), IM, on Day 29.
  Interventions: Biological: Norovirus GI.1/GII.4 Bivalent VLP Vaccine; Drug: 0.9% sodium chloride (saline)

INTERVENTIONS:
Biological: Norovirus GI.1/GII.4 Bivalent VLP Vaccine — Norovirus GI.1/GII.4 bivalent VLP vaccine adjuvanted with aluminum hydroxide, without MPL for IM injection
  Arms: Arm 1: NoV Vaccine Formulation A _1-Dose; Arm 2: NoV Vaccine Formulation A _2-Dose; Arm 5: NoV Vaccine Formulation A_1-Dose
Drug: 0.9% sodium chloride (saline) — norovirus bivalent placebo-matching vaccine
  Arms: Arm 1: NoV Vaccine Formulation A _1-Dose; Arm 3: NoV Vaccine Formulation B_1-Dose; Arm 5: NoV Vaccine Formulation A_1-Dose
Biological: Norovirus GI.1/GII.4 Bivalent VLP Vaccine — Norovirus GI.1/GII.4 bivalent VLP vaccine adjuvanted with MPL and aluminum hydroxide for IM injection
  Arms: Arm 3: NoV Vaccine Formulation B_1-Dose; Arm 4: NoV Vaccine Formulation B_2-Dose

SUMMARY:
The purpose of this study is to further develop a formulation and dose regimen of the norovirus GI.1/GII.4 bivalent virus-like particle (VLP) vaccine that is immunogenic and safe in an elderly population aged 60 years and above.

DETAILED DESCRIPTION:
The vaccine being tested in this study is called norovirus GI.1/GII.4 bivalent virus-like particle (VLP) vaccine adjuvanted with aluminum hydroxide (Formulation A) or adjuvanted with monophosphoryl lipid A (MPL) and aluminum hydroxide (Formulation B). Two norovirus vaccine formulations are being tested to select for further development the formulation that will generate an optimal specific antibody response that may provide protection against norovirus and is safe in a population aged 60 years and above. This study will look at side effects and the level of antibodies to norovirus formed in people who will be injected with different formulations of the norovirus vaccine candidate.

The study will enroll approximately 325 patients. Participants will be randomly assigned (by chance) to one of five treatment groups.

* Norovirus GI.1/GII.4 bivalent VLP vaccine (Formulation A) 1-dose, participants ≥ 60 years
* Norovirus GI.1/GII.4 bivalent VLP vaccine (Formulation A) 2-dose, participants ≥ 60 years
* Norovirus GI.1/GII.4 bivalent VLP vaccine (Formulation B) 1-dose, participants ≥ 60 years
* Norovirus GI.1/GII.4 bivalent VLP vaccine (Formulation B) 2-dose, participants ≥ 60 years
* Norovirus GI.1/GII.4 bivalent VLP vaccine (Formulation A) 1-dose, participants 18 to 49 years All participants in the age of 60 years and older will be administered either NoV vaccine (Formulation A or B) or placebo on Day 1 and NoV vaccine (Formulation A or B) on Day 29 of the study. In order to keep the treatment arms undisclosed to the patient and the doctor, those randomized to the one dose groups will receive a dose of placebo (this is a saline solution that has no active ingredient) on Day 1 followed by the NoV vaccine on Day 29. Those randomized to 2 doses with receive the NoV vaccine on Day 1 and Day 29. In case of an urgent medical need a participant can be unblinded.

Adults aged 18 to 49 will receive placebo on Day 1 followed by NoV vaccine Formulation A on Day 29.

Participants will be asked to record any reactions/ symptoms that may be related or not to the vaccine in a diary card for 28 days after each vaccination.

This multi-center trial will be conducted in the United States of America. The overall time to participate in this study is up to 393 days. Participants will make multiple visits to the clinic including a final follow-up visit on Day 393.

ELIGIBILITY:
Inclusion Criteria:

1. Is aged 18 to 49 years, or 60 years and older at the time of enrollment;
2. Participants who are in good health, or in stable health status with no exclusionary medical or neuropsychiatric conditions at the time of entry into the trial as determined by medical history, physical examination (including vital signs) and clinical judgment of the Investigator;
3. Participant signs and dates a written, Informed Consent Form (ICF) and any required privacy authorization prior to the initiation of any trial procedures, after the nature of the trial has been explained according to local regulatory requirements;
4. Participants who can comply with trial procedures and are available for the duration of follow-up.

Exclusion Criteria:

1. Has a known hypersensitivity or allergy to any of the Norovirus (NoV) GI.1/GII.4 Bivalent virus-like particle (VLP) Vaccine components;
2. Has a clinically significant active infection (as assessed by the Investigator) or body temperature ≥38°C/100.4°F within 3 days of the intended date of vaccination;
3. Participants with the presence of significant acute or chronic, uncontrolled medical or neuropsychiatric illness. Uncontrolled was defined as:

   Requiring institution of new medical or surgical treatment within 3 months prior to immunization, or Requiring a change in medication dosage in the 3 months prior to immunization due to uncontrolled symptoms or drug toxicity (elective dosage adjustments in stable participants were acceptable), or Hospitalization or an event fulfilling the definition of a serious adverse event within 3 months prior immunization.
4. Has any unstable medical or neuropsychiatric condition, which in the Investigator's opinion poses a risk of unusual magnitude for the participant's age group of hospitalization, death, or an event meeting the definition of a serious adverse event within 2 months of immunization. The intent of this criterion is to recognize and allow for the frequent existence of significant health concerns in this population; but exclude those participants who are experiencing an acute decline in health status;
5. Has any medical or neuropsychiatric condition, which in the Investigator's opinion, rendered the participant incompetent to provide informed consent or unable to provide valid safety observations and reports;
6. Has behavioral or cognitive impairment or psychiatric disease that, in the opinion of the Investigator, may interfere with the participant's ability to participate in the trial;
7. Participants with any history of progressive or severe neurologic disorder, history of seizure, or history of neuro-inflammatory disease (e.g. Guillain-Barre syndrome);
8. Participants with history or any illness that, in the opinion of the Investigator, might interfere with the results of the trial or pose additional risk to the participants due to participation in the trial;
9. Has known or suspected autoimmune disease;
10. Has known or suspected impairment/alteration of immune function, including:

    Chronic use of oral steroids (Equivalent to 20 mg/day prednisone ≥ 12 weeks/≥ 2 mg/kg body weight/day prednisone ≥ 2 weeks) within 60 days prior to Day 1 (use of inhaled, intranasal, or topical corticosteroids is allowed).

    Receipt of parenteral steroids (Equivalent to 20 mg/day prednisone ≥ 12 weeks/≥ 2 mg/kg body weight/day prednisone ≥ 2 weeks) within 60 days prior to Day 1.

    Receipt of immunosuppressive therapy within 3 months prior to Day 1. Receipt of immunostimulants within 60 days prior to Day 1. Receipt of parenteral, epidural or intra-articular immunoglobulin preparation, blood products, and/or plasma derivatives within 3 months prior to Day 1 or planned during the full length of the trial.

    Human Immunodeficiency Virus (HIV) infection or HIV-related disease. Genetic immunodeficiency.
11. Has abnormalities of splenic or thymic function;
12. Has any significant disorder of coagulation or treatment with anticoagulant therapy that would increase the risk of intramuscular (IM) injection. Persons receiving prophylactic antiplatelet medication such as low dose of acetylsalicylic acid are eligible;
13. Has any serious chronic or progressive disease according to judgment of the Investigator: cancer (malignancy other than resolved/excised skin lesion), insulin dependent Type I diabetes (Type II diabetes is accepted), cardiac, renal or hepatic disease;
14. Has body mass index (BMI) greater than or equal to 35 kg/m^2 (= weight in kg/[height in meters^2]);
15. Is participating in any clinical trial with another investigational product 30 days prior to first trial visit or intent to participate in another clinical trial at any time during the conduct of this trial;
16. Participants who received any other vaccines within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to enrollment in this trial or who are planning to receive any vaccine within 28 days of investigational vaccine administration;
17. Participants involved in trial conduct or their first degree relatives;
18. Has history of substance or alcohol abuse within the past 2 years;
19. Females who are pregnant or breastfeeding;
20. If female of childbearing potential, sexually active with a male partner who has not been sterilized, and has not used any of the "acceptable contraceptive methods" for at least 2 months prior to trial entry:

    Of childbearing potential is defined as status post onset of menarche and not meeting any of the following conditions: menopausal for at least 2 years, status after bilateral tubal ligation for at least 1 year, status after bilateral oophorectomy, or status after hysterectomy.

    Acceptable birth control methods are defined as one or more of the following: i. Hormonal contraceptive (such as oral, injection, transdermal patch, implant, cervical ring); ii. Barrier (condom with spermicide or diaphragm with spermicide) each and every time during intercourse; iii. Intrauterine device (IUD); iv. Monogamous relationship with vasectomized partner. Partner must have been vasectomized for at least six months prior to the participants' trial entry.
21. If female of childbearing potential and sexually active, refusal to use an "acceptable contraceptive method" from Day 1 and throughout the duration of the trial. In addition, they must be advised not to donate ova during this period;
22. Females with any positive or indeterminate pregnancy test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2016-10-28 (Actual); Study Completion 2017-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (10):
- United States (10):
  - Simon Williamson Clinic, Birmingham, Alabama
  - Fountain Hills Family Practice, P.C., Fountain Hills, Arizona
  - Southwest Family Medicine, Littleton, Colorado
  - Miami Research Associates, Miami, Florida
  - Johnson County Clin-Trials, Lenexa, Kansas
  - St. Louis University, School of Medicine, St Louis, Missouri
  - Regional Clinical Research Inc., Endwell, New York
  - University of Rochester, Rochester, New York
  - Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio
  - Group Health Research Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 10 investigative sites in United States from 1 February 2016 to 31 October 2017.
Pre-assignment Details: Healthy elderly volunteers were enrolled and randomized in 1:1:1:1 ratio in 4 arm groups to receive either one or two doses of one of the 2 formulations (A or B) of norovirus (NoV) GI.1/GII4 bivalent virus like particle (VLP) vaccine or placebo. Healthy young adults received both placebo and formulation A.
Groups:
- Arm 1: NoV Vaccine Formulation A_1-Dose: Participants ≥ 60 years of age, 1-dose regimen: Norovirus bivalent placebo-matching vaccine, intramuscularly (IM), on Day 1, followed by norovirus (NoV) GI.1 (15 μg)/GII.4 (50 μg) bivalent virus-like particle (VLP) vaccine (Formulation A), IM, on Day 29.
- Arm 2: NoV Vaccine Formulation A_2-Dose: Participants ≥ 60 years of age, 2-dose regimen: Norovirus GI.1 (15 μg)/GII.4 (50 μg) bivalent VLP vaccine (Formulation A), IM, on Days 1 and 29.
Period: Overall Study
Arm/Group | Arm 1: NoV Vaccine Formulation A_1-Dose | Arm 2: NoV Vaccine Formulation A_2-Dose | Arm 3: NoV Vaccine Formulation B_1-Dose | Arm 4: NoV Vaccine Formulation B_2-Dose | Arm 5: NoV Vaccine Formulation A_1-Dose
Started | 76 | 74 | 72 | 72 | 26
Completed | 73 | 72 | 70 | 71 | 23
Not Completed | 3 | 2 | 2 | 1 | 3
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 2 | 0 | 2 | 0 | 0
Not completed — Death | 1 | 1 | 0 | 1 | 0
Not completed — Reason not Specified | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomized Set included all randomized participants regardless of whether any study vaccine (NoV VLP vaccine or placebo) was received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: NoV Vaccine Formulation A_1-Dose | Arm 2: NoV Vaccine Formulation A_2-Dose | Arm 3: NoV Vaccine Formulation B_1-Dose | Arm 4: NoV Vaccine Formulation B_2-Dose | Arm 5: NoV Vaccine Formulation A_1-Dose | Total
Number analyzed (Participants) | 76 | 74 | 72 | 72 | 26 | 320
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Data is reported for elderly participants only.
  years
    number analyzed (Participants) | 76 | 74 | 72 | 72 | 0 | 294
    (all) | 78.0 (9.14) | 77.4 (9.32) | 76.7 (9.22) | 77.7 (9.07) |  | 77.4 (9.15)
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Data is reported for young adult participants only.
  years
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 26 | 26
    (all) |  |  |  |  | 34.6 (8.46) | 34.6 (8.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 41 | 40 | 40 | 16 | 181
  Male | 32 | 33 | 32 | 32 | 10 | 139
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 3 | 4 | 2 | 19
  Not Hispanic or Latino | 72 | 68 | 69 | 68 | 24 | 301
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 1 | 2 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1 | 2
  Black or African American | 2 | 5 | 2 | 0 | 2 | 11
  White | 72 | 69 | 68 | 70 | 20 | 299
  More than one race | 0 | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 76 | 74 | 72 | 72 | 26 | 320
Height [Mean (Standard Deviation); unit: cm] — Population: Data is reported for elderly participants only.
  cm
    number analyzed (Participants) | 76 | 74 | 72 | 72 | 0 | 294
    (all) | 166.8 (9.95) | 167.3 (9.52) | 168.0 (9.17) | 167.4 (10.26) |  | 167.3 (9.69)
Height [Mean (Standard Deviation); unit: cm] — Population: Data is reported for young adult participants only for whom data for height was available at Baseline.
  cm
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 25 | 25
    (all) |  |  |  |  | 169.4 (11.42) | 169.4 (11.42)
Weight [Mean (Standard Deviation); unit: kg] — Population: Data is reported for elderly participants only.
  kg
    number analyzed (Participants) | 76 | 74 | 72 | 72 | 0 | 294
    (all) | 75.56 (14.376) | 73.76 (13.804) | 77.26 (14.404) | 74.34 (13.965) |  | 75.22 (14.131)
Weight [Mean (Standard Deviation); unit: kg] — Population: Data is reported for young adult participants only for whom data for weight was available at Baseline.
  kg
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 25 | 25
    (all) |  |  |  |  | 78.22 (15.357) | 78.22 (15.357)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI=Weight (kg)/height (m^2) Population: Data is reported for elderly participants only.
  kg/m^2
    number analyzed (Participants) | 76 | 74 | 72 | 72 | 0 | 294
    (all) | 27.01 (3.554) | 26.28 (3.958) | 27.29 (3.899) | 26.46 (3.909) |  | 26.76 (3.833)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI=Weight (kg)/height (m^2) Population: Data is reported for young adult participants only for whom data for BMI was available at Baseline.
  kg/m^2
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 25 | 25
    (all) |  |  |  |  | 27.22 (4.481) | 27.22 (4.481)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a 4-Fold Rise or Greater in Serum Anti-norovirus Antibody Titers for Both GI.1 and GII.4 Virus Like Particles (VLP) as Measured by Histoblood Group Antigen (HBGA) Blocking Assay on Day 57
Time Frame: Day 57
Population: Per Protocol Set (PPS) included all participants in the Full Analysis Set (FAS), who receive the planned vaccination [both doses of vaccine, i.e. Norovirus (NoV) VLP vaccine or placebo], and did not have major protocol violations. Overall number of participants analyzed is the number of participants with data available for analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1: NoV Vaccine Formulation A_1-Dose | Arm 2: NoV Vaccine Formulation A_2-Dose | Arm 3: NoV Vaccine Formulation B_1-Dose | Arm 4: NoV Vaccine Formulation B_2-Dose | Arm 5: NoV Vaccine Formulation A_1-Dose
Number analyzed (Participants) | 71 | 65 | 62 | 66 | 24
percentage of participants | 42.3 [30.6 to 54.6] | 41.5 [29.4 to 54.4] | 56.5 [43.3 to 69.0] | 63.6 [50.9 to 75.1] | 45.8 [25.6 to 67.2]

2. Primary Outcome: Percentage of Participants With Solicited Local Adverse Events (AEs) at Injection Site for 7-day Period (Including Day of Vaccination) After First Vaccination on Day 1
Description: Solicited local AEs at the injection site that occurred within 7 days after each vaccination were collected using a diary and included pain, erythema swelling and induration.
Time Frame: Within 7 days of first vaccination on Day 1
Population: Safety Analysis Set (SAF) included all participants who received at least 1 dose of vaccine (NoV VLP vaccine or placebo). Number analyzed is the number of participants with evaluable data for the specific category.
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: NoV Vaccine Formulation A_1-Dose | Arm 2: NoV Vaccine Formulation A_2-Dose | Arm 3: NoV Vaccine Formulation B_1-Dose | Arm 4: NoV Vaccine Formulation B_2-Dose | Arm 5: NoV Vaccine Formulation A_1-Dose
Number analyzed (Participants) | 76 | 74 | 72 | 72 | 25
percentage of participants
  Any Solicited Local AEs: number analyzed (Participants) | 76 | 73 | 72 | 72 | 25
  Any Solicited Local AEs | 6.6 | 26.0 | 15.3 | 34.7 | 4.0
  Pain: number analyzed (Participants) | 76 | 73 | 72 | 72 | 25
  Pain | 5.3 | 23.3 | 9.7 | 34.7 | 4.0
  Erythema: number analyzed (Participants) | 76 | 73 | 72 | 72 | 25
  Erythema | 1.3 | 2.7 | 4.2 | 1.4 | 4.0
  Swelling: number analyzed (Participants) | 76 | 73 | 72 | 72 | 25
  Swelling | 0.0 | 2.7 | 2.8 | 1.4 | 0.0
  Induration: number analyzed (Participants) | 76 | 73 | 72 | 72 | 25
  Induration | 0.0 | 1.4 | 1.4 | 1.4 | 0.0

3. Primary Outcome: Percentage of Participants With Solicited Local Adverse Events (AEs) at Injection Site for 7-day Period (Including Day of Vaccination) After Second Vaccination on Day 29
Description: Solicited local AEs at the injection site that occurred within 7 days after each vaccination were collected using a diary and included pain, erythema, swelling and induration.
Time Frame: Within 7 days of second vaccination on Day 29
Population: SAF included all participants who received at least 1 dose of vaccine (NoV VLP vaccine or placebo). Overall number of participants analyzed is the number of participants with data available for analyses.
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: NoV Vaccine Formulation A_1-Dose | Arm 2: NoV Vaccine Formulation A_2-Dose | Arm 3: NoV Vaccine Formulation B_1-Dose | Arm 4: NoV Vaccine Formulation B_2-Dose | Arm 5: NoV Vaccine Formulation A_1-Dose
Number analyzed (Participants) | 73 | 69 | 68 | 66 | 24
percentage of participants
  Any Solicited Local AEs | 37.0 | 21.7 | 38.2 | 39.4 | 41.7
  Pain | 32.9 | 21.7 | 38.2 | 37.9 | 41.7
  Erythema | 2.7 | 0.0 | 1.5 | 3.0 | 0.0
  Swelling | 1.4 | 0.0 | 1.5 | 1.5 | 0.0
  Induration | 1.4 | 0.0 | 1.5 | 1.5 | 0.0

4. Primary Outcome: Percentage of Participants With Solicited Systemic Adverse Events (AEs) for 7-day Period (Including Day of Vaccination) After First Vaccination on Day 1
Description: Solicited systemic AEs that occurred within 7 days after each vaccination were collected using a diary and included headache, fatigue, myalgia, arthralgia, vomiting, and diarrhea.
Time Frame: Within 7 days of first vaccination on Day 1
Population: SAF included all participants who received at least 1 dose of vaccine (NoV VLP vaccine or placebo). Number analyzed is the number of participants with evaluable data for the specific category.
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: NoV Vaccine Formulation A_1-Dose | Arm 2: NoV Vaccine Formulation A_2-Dose | Arm 3: NoV Vaccine Formulation B_1-Dose | Arm 4: NoV Vaccine Formulation B_2-Dose | Arm 5: NoV Vaccine Formulation A_1-Dose
Number analyzed (Participants) | 76 | 74 | 72 | 72 | 25
percentage of participants
  Any solicited systemic AEs: number analyzed (Participants) | 76 | 73 | 72 | 72 | 25
  Any solicited systemic AEs | 28.9 | 34.2 | 30.6 | 44.4 | 36.0
  Headache: number analyzed (Participants) | 76 | 73 | 72 | 72 | 25
  Headache | 7.9 | 2.7 | 11.1 | 12.5 | 20.0
  Fatigue: number analyzed (Participants) | 76 | 73 | 72 | 72 | 25
  Fatigue | 18.4 | 24.7 | 9.7 | 27.8 | 28.0
  Myalgia: number analyzed (Participants) | 76 | 73 | 72 | 72 | 25
  Myalgia | 5.3 | 13.7 | 11.1 | 20.8 | 16.0
  Arthralgia: number analyzed (Participants) | 76 | 73 | 72 | 72 | 25
  Arthralgia | 5.3 | 8.2 | 6.9 | 6.9 | 4.0
  Vomiting: number analyzed (Participants) | 76 | 73 | 72 | 72 | 25
  Vomiting | 0.0 | 1.4 | 0.0 | 2.8 | 0.0
  Diarrhea: number analyzed (Participants) | 76 | 73 | 72 | 72 | 25
  Diarrhea | 5.3 | 6.8 | 8.3 | 18.1 | 8.0

5. Primary Outcome: Percentage of Participants With Solicited Systemic Adverse Events (AEs) for 7-day Period (Including Day of Vaccination) After Second Vaccination on Day 29
Description: as for outcome 4
Time Frame: Within 7 days of second vaccination on Day 29
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: NoV Vaccine Formulation A_1-Dose | Arm 2: NoV Vaccine Formulation A_2-Dose | Arm 3: NoV Vaccine Formulation B_1-Dose | Arm 4: NoV Vaccine Formulation B_2-Dose | Arm 5: NoV Vaccine Formulation A_1-Dose
Number analyzed (Participants) | 73 | 69 | 68 | 66 | 24
percentage of participants
  Any solicited systemic AEs | 19.2 | 20.3 | 20.6 | 28.8 | 16.7
  Headache | 8.2 | 5.8 | 5.9 | 6.1 | 4.2
  Fatigue | 12.3 | 15.9 | 13.2 | 15.2 | 8.3
  Myalgia | 6.8 | 5.8 | 7.4 | 13.6 | 4.2
  Arthralgia | 4.1 | 7.2 | 4.4 | 6.1 | 4.2
  Vomiting | 0.0 | 0.0 | 0.0 | 1.5 | 0.0
  Diarrhea | 1.4 | 4.3 | 2.9 | 4.5 | 0.0

6. Primary Outcome: Percentage of Participants With Elevated Body Temperature ≥38°C (Defined as Fever) for 7-day Period (Including Day of Vaccination) After First Vaccination on Day 1
Description: The body temperature measurement was performed using the thermometer for 7 days after each vaccination. The highest body temperature observed each day was recorded on the diary card. An elevated temperature is ≥ 38 °C or 100.4°F (considered as fever).
Time Frame: Within 7 days of first vaccination on Day 1
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: NoV Vaccine Formulation A_1-Dose | Arm 2: NoV Vaccine Formulation A_2-Dose | Arm 3: NoV Vaccine Formulation B_1-Dose | Arm 4: NoV Vaccine Formulation B_2-Dose | Arm 5: NoV Vaccine Formulation A_1-Dose
Number analyzed (Participants) | 76 | 72 | 72 | 71 | 25
percentage of participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

7. Primary Outcome: Percentage of Participants With Elevated Body Temperature ≥38°C (Defined as Fever) for 7-day Period (Including Day of Vaccination) After Second Vaccination on Day 29
Description: as for outcome 6
Time Frame: Within 7 days of second vaccination on Day 29
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: NoV Vaccine Formulation A_1-Dose | Arm 2: NoV Vaccine Formulation A_2-Dose | Arm 3: NoV Vaccine Formulation B_1-Dose | Arm 4: NoV Vaccine Formulation B_2-Dose | Arm 5: NoV Vaccine Formulation A_1-Dose
Number analyzed (Participants) | 73 | 69 | 68 | 66 | 24
percentage of participants | 0.0 | 0.0 | 0.0 | 1.5 | 0.0

8. Primary Outcome: Percentage of Participants With At Least One Unsolicited Adverse Event (AE) Within 28-days After First Vaccination on Day 1
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment.
Time Frame: Within 28 days of first vaccination on Day 1
Population: SAF included all participants who received at least 1 dose of vaccine (NoV VLP vaccine or placebo).
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: NoV Vaccine Formulation A_1-Dose | Arm 2: NoV Vaccine Formulation A_2-Dose | Arm 3: NoV Vaccine Formulation B_1-Dose | Arm 4: NoV Vaccine Formulation B_2-Dose | Arm 5: NoV Vaccine Formulation A_1-Dose
Number analyzed (Participants) | 76 | 74 | 72 | 72 | 25
percentage of participants | 32.9 | 28.4 | 33.3 | 26.4 | 20.0

9. Primary Outcome: Percentage of Participants With At Least One Unsolicited Adverse Event (AE) Within 28-days After Second Vaccination on Day 29
Description: as for outcome 8
Time Frame: Within 28 days of second vaccination on Day 29
Population: SAF included all participants who received at least 1 dose of vaccine (NoV VLP vaccine or placebo). Overall number of participants analyzed is number of participants with data available for analyses.
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: NoV Vaccine Formulation A_1-Dose | Arm 2: NoV Vaccine Formulation A_2-Dose | Arm 3: NoV Vaccine Formulation B_1-Dose | Arm 4: NoV Vaccine Formulation B_2-Dose | Arm 5: NoV Vaccine Formulation A_1-Dose
Number analyzed (Participants) | 73 | 69 | 68 | 66 | 24
percentage of participants | 34.2 | 18.8 | 25.0 | 30.3 | 8.3

10. Primary Outcome: Percentage of Participants With At Least One Serious Adverse Event (SAE)
Description: An SAE is any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically important due to other reasons than the above mentioned criteria.
Time Frame: From first vaccination up to Day 393
Population: SAF included all participants who received at least 1 dose of vaccine (NoV VLP vaccine or placebo).
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: NoV Vaccine Formulation A_1-Dose | Arm 2: NoV Vaccine Formulation A_2-Dose | Arm 3: NoV Vaccine Formulation B_1-Dose | Arm 4: NoV Vaccine Formulation B_2-Dose | Arm 5: NoV Vaccine Formulation A_1-Dose
Number analyzed (Participants) | 76 | 74 | 72 | 72 | 25
percentage of participants | 9.2 | 12.2 | 23.6 | 12.5 | 0.0

11. Secondary Outcome: Percentage of Participants With a 4-Fold Rise or Greater in Serum Anti-norovirus Antibody Titers for Both GI.1 VLP and GII.4 VLP as Measured by HBGA Blocking Assay
Time Frame: Days 8, 29, 36, 211 and 393
Population: PPS included all participants in the FAS, who received the planned vaccination (both doses of vaccine, i.e. NoV VLP vaccine or placebo), and did not have major protocol violations. Number analyzed is the number of participants with evaluable data at the given time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1: NoV Vaccine Formulation A_1-Dose | Arm 2: NoV Vaccine Formulation A_2-Dose | Arm 3: NoV Vaccine Formulation B_1-Dose | Arm 4: NoV Vaccine Formulation B_2-Dose | Arm 5: NoV Vaccine Formulation A_1-Dose
Number analyzed (Participants) | 72 | 67 | 66 | 66 | 24
percentage of participants
  Day 8: number analyzed (Participants) | 72 | 65 | 66 | 65 | 23
  Day 8 | 0.0 [0.0 to 5.0] | 33.8 [22.6 to 46.6] | 0.0 [0.0 to 5.4] | 55.4 [42.5 to 67.7] | 0.0 [0.0 to 14.8]
  Day 29: number analyzed (Participants) | 72 | 66 | 66 | 66 | 24
  Day 29 | 0.0 [0.0 to 5.0] | 40.9 [29.0 to 53.7] | 0.0 [0.0 to 5.4] | 54.5 [41.8 to 66.9] | 0.0 [0.0 to 14.2]
  Day 36: number analyzed (Participants) | 72 | 66 | 64 | 66 | 23
  Day 36 | 26.4 [16.7 to 38.1] | 45.5 [33.1 to 58.2] | 34.4 [22.9 to 47.3] | 63.6 [50.9 to 75.1] | 43.5 [23.2 to 65.5]
  Day 211: number analyzed (Participants) | 71 | 66 | 64 | 66 | 23
  Day 211 | 15.5 [8.0 to 26.0] | 18.2 [9.8 to 29.6] | 28.1 [17.6 to 40.8] | 30.3 [19.6 to 42.9] | 8.7 [1.1 to 28.0]
  Day 393: number analyzed (Participants) | 70 | 64 | 63 | 65 | 23
  Day 393 | 12.9 [6.1 to 23.0] | 10.9 [4.5 to 21.2] | 19.0 [10.2 to 30.9] | 16.9 [8.8 to 28.3] | 13.0 [2.8 to 33.6]

12. Secondary Outcome: Percentage of Participants With a 4-Fold Rise or Greater in Serum Anti-norovirus GI.1 VLP Antibody Titers (HBGA)
Time Frame: Days 8, 29, 36, 57, 211 and 393
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1: NoV Vaccine Formulation A_1-Dose | Arm 2: NoV Vaccine Formulation A_2-Dose | Arm 3: NoV Vaccine Formulation B_1-Dose | Arm 4: NoV Vaccine Formulation B_2-Dose | Arm 5: NoV Vaccine Formulation A_1-Dose
Number analyzed (Participants) | 72 | 67 | 66 | 66 | 24
percentage of participants
  Day 8: number analyzed (Participants) | 72 | 65 | 66 | 65 | 23
  Day 8 | 1.4 [0.0 to 7.5] | 63.1 [50.2 to 74.7] | 0.0 [0.0 to 5.4] | 76.9 [64.8 to 86.5] | 0.0 [0.0 to 14.8]
  Day 29: number analyzed (Participants) | 72 | 66 | 66 | 66 | 24
  Day 29 | 0.0 [0.0 to 5.0] | 72.7 [60.4 to 83.0] | 0.0 [0.0 to 5.4] | 77.3 [65.3 to 86.7] | 0.0 [0.0 to 14.2]
  Day 36: number analyzed (Participants) | 72 | 66 | 64 | 66 | 23
  Day 36 | 55.6 [43.4 to 67.3] | 74.2 [62.0 to 84.2] | 65.6 [52.7 to 77.1] | 89.4 [79.4 to 95.6] | 60.9 [38.5 to 80.3]
  Day 57: number analyzed (Participants) | 71 | 65 | 62 | 66 | 24
  Day 57 | 64.8 [52.5 to 75.8] | 80.0 [68.2 to 88.9] | 74.2 [61.5 to 84.5] | 89.4 [79.4 to 95.6] | 62.5 [40.6 to 81.2]
  Day 211: number analyzed (Participants) | 71 | 66 | 64 | 66 | 23
  Day 211 | 33.8 [23.0 to 46.0] | 57.6 [44.8 to 69.7] | 54.7 [41.7 to 67.2] | 57.6 [44.8 to 69.7] | 26.1 [10.2 to 48.4]
  Day 393: number analyzed (Participants) | 70 | 64 | 63 | 65 | 23
  Day 393 | 25.7 [16.0 to 37.6] | 50.0 [37.2 to 62.8] | 41.3 [29.0 to 54.4] | 47.7 [35.1 to 60.5] | 30.4 [13.2 to 52.9]

13. Secondary Outcome: Percentage of Participants With a 4-Fold Rise or Greater in Serum Anti-norovirus GII.4 VLP Antibody Titers (HBGA)
Time Frame: Days 8, 29, 36, 57, 211 and 393
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1: NoV Vaccine Formulation A_1-Dose | Arm 2: NoV Vaccine Formulation A_2-Dose | Arm 3: NoV Vaccine Formulation B_1-Dose | Arm 4: NoV Vaccine Formulation B_2-Dose | Arm 5: NoV Vaccine Formulation A_1-Dose
Number analyzed (Participants) | 72 | 67 | 66 | 66 | 24
percentage of participants
  Day 8: number analyzed (Participants) | 72 | 66 | 66 | 65 | 23
  Day 8 | 0.0 [0.0 to 5.0] | 54.5 [41.8 to 66.9] | 1.5 [0.0 to 8.2] | 69.2 [56.6 to 80.1] | 0.0 [0.0 to 14.8]
  Day 29 | 1.4 [0.0 to 7.5] | 59.7 [47.0 to 71.5] | 0.0 [0.0 to 5.4] | 71.2 [58.7 to 81.7] | 0.0 [0.0 to 14.2]
  Day 36: number analyzed (Participants) | 72 | 67 | 64 | 66 | 23
  Day 36 | 56.9 [44.7 to 68.6] | 62.7 [50.0 to 74.2] | 53.1 [40.2 to 65.7] | 71.2 [58.7 to 81.7] | 78.3 [56.3 to 92.5]
  Day 57: number analyzed (Participants) | 71 | 66 | 62 | 66 | 24
  Day 57 | 67.6 [55.5 to 78.2] | 57.6 [44.8 to 69.7] | 74.2 [61.5 to 84.5] | 71.2 [58.7 to 81.7] | 66.7 [44.7 to 84.4]
  Day 211: number analyzed (Participants) | 71 | 66 | 64 | 66 | 23
  Day 211 | 39.4 [28.0 to 51.7] | 34.8 [23.5 to 47.6] | 45.3 [32.8 to 58.3] | 45.5 [33.1 to 58.2] | 47.8 [26.8 to 69.4]
  Day 393: number analyzed (Participants) | 70 | 65 | 63 | 65 | 23
  Day 393 | 34.3 [23.3 to 46.6] | 30.8 [19.9 to 43.4] | 33.3 [22.0 to 46.3] | 36.9 [25.3 to 49.8] | 39.1 [19.7 to 61.5]

14. Secondary Outcome: Geometric Mean Titer (GMT) GI.1 VLP Antibody Titers (HBGA)
Description: GMT GI.1 VLP antibody titers measured by HBGA blocking assay are reported.
Time Frame: Baseline (Day 1), Days 8, 29, 36, 57, 211 and 393
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Arm 1: NoV Vaccine Formulation A_1-Dose | Arm 2: NoV Vaccine Formulation A_2-Dose | Arm 3: NoV Vaccine Formulation B_1-Dose | Arm 4: NoV Vaccine Formulation B_2-Dose | Arm 5: NoV Vaccine Formulation A_1-Dose
Number analyzed (Participants) | 72 | 67 | 66 | 66 | 24
titer
  Baseline (Day 1): number analyzed (Participants) | 72 | 66 | 66 | 66 | 24
  Baseline (Day 1) | 26.5 [20.9 to 33.6] | 29.0 [22.3 to 37.7] | 26.7 [20.9 to 34.2] | 23.9 [19.8 to 28.8] | 22.0 [15.4 to 31.6]
  Day 8: number analyzed (Participants) | 72 | 66 | 66 | 65 | 23
  Day 8 | 26.6 [20.9 to 33.9] | 282.4 [193.2 to 412.6] | 26.5 [20.9 to 33.6] | 332.3 [209.9 to 526.1] | 21.7 [15.3 to 30.8]
  Day 29 | 26.2 [20.8 to 33.0] | 373.6 [266.9 to 523.0] | 27.3 [21.4 to 34.8] | 285.5 [192.9 to 422.6] | 21.7 [15.3 to 30.9]
  Day 36: number analyzed (Participants) | 72 | 67 | 64 | 66 | 23
  Day 36 | 194.2 [130.3 to 289.4] | 361.1 [266.5 to 489.2] | 280.1 [184.3 to 425.7] | 338.9 [247.7 to 463.7] | 150.8 [75.0 to 303.4]
  Day 57: number analyzed (Participants) | 71 | 66 | 62 | 66 | 24
  Day 57 | 177.0 [124.4 to 251.9] | 353.6 [268.6 to 465.6] | 262.2 [180.5 to 381.0] | 317.1 [238.3 to 421.9] | 117.7 [63.1 to 219.5]
  Day 211: number analyzed (Participants) | 71 | 66 | 64 | 66 | 23
  Day 211 | 81.8 [60.4 to 110.6] | 160.5 [116.5 to 221.1] | 128.3 [92.7 to 177.7] | 126.7 [92.7 to 173.3] | 54.1 [30.1 to 97.0]
  Day 393: number analyzed (Participants) | 70 | 65 | 63 | 65 | 23
  Day 393 | 60.2 [43.9 to 82.5] | 112.2 [80.4 to 156.5] | 85.7 [61.8 to 118.9] | 84.6 [60.3 to 118.5] | 41.0 [23.3 to 72.2]

15. Secondary Outcome: GMT of Anti-norovirus GII.4 VLP Antibody Titers (HBGA)
Description: GMT of anti-norovirus GII.4 VLP antibody titers measured by HBGA blocking assay are reported.
Time Frame: Baseline (Day 1), Days 8, 29, 36, 57, 211 and 393
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Arm 1: NoV Vaccine Formulation A_1-Dose | Arm 2: NoV Vaccine Formulation A_2-Dose | Arm 3: NoV Vaccine Formulation B_1-Dose | Arm 4: NoV Vaccine Formulation B_2-Dose | Arm 5: NoV Vaccine Formulation A_1-Dose
Number analyzed (Participants) | 72 | 67 | 66 | 66 | 24
titer
  Baseline (Day 1) | 66.5 [48.4 to 91.4] | 100.3 [70.8 to 142.2] | 99.5 [67.4 to 146.8] | 86.1 [60.7 to 122.2] | 78.7 [43.7 to 141.4]
  Day 8: number analyzed (Participants) | 72 | 66 | 66 | 65 | 23
  Day 8 | 60.7 [43.8 to 84.2] | 694.9 [462.6 to 1043.9] | 94.1 [65.2 to 135.8] | 994.9 [724.8 to 1365.8] | 75.2 [41.3 to 137.0]
  Day 29 | 58.6 [42.0 to 81.6] | 787.7 [524.9 to 1182.1] | 82.8 [57.5 to 119.3] | 876.1 [648.5 to 1183.6] | 67.2 [38.0 to 118.8]
  Day 36: number analyzed (Participants) | 72 | 67 | 64 | 66 | 23
  Day 36 | 556.5 [354.6 to 873.2] | 757.1 [526.7 to 1088.4] | 733.8 [460.0 to 1170.7] | 799.4 [604.1 to 1057.9] | 1234.5 [627.3 to 2429.4]
  Day 57: number analyzed (Participants) | 71 | 66 | 62 | 66 | 24
  Day 57 | 528.0 [366.2 to 761.2] | 600.6 [417.3 to 864.5] | 790.8 [543.4 to 1151.0] | 613.6 [475.5 to 791.8] | 742.0 [406.9 to 1352.9]
  Day 211: number analyzed (Participants) | 71 | 66 | 64 | 66 | 23
  Day 211 | 222.0 [158.2 to 311.6] | 298.9 [204.6 to 436.6] | 318.6 [228.6 to 444.1] | 315.9 [233.7 to 427.1] | 280.3 [163.4 to 480.8]
  Day 393: number analyzed (Participants) | 70 | 65 | 63 | 65 | 23
  Day 393 | 188.9 [129.7 to 275.1] | 249.8 [164.4 to 379.8] | 265.9 [184.4 to 383.6] | 278.9 [204.9 to 379.7] | 223.4 [114.5 to 436.0]

16. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of Anti-norovirus GI.1 VLP Antibody Titers (HBGA)
Description: GMFR of anti-norovirus GI.1 VLP antibody titers measured by HBGA blocking assay are reported. The fold rise was calculated as the ratio of the post-vaccination titer level to the pre-vaccination titer level.
Time Frame: Days 8, 29, 36, 57, 211 and 393
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Arm 1: NoV Vaccine Formulation A_1-Dose | Arm 2: NoV Vaccine Formulation A_2-Dose | Arm 3: NoV Vaccine Formulation B_1-Dose | Arm 4: NoV Vaccine Formulation B_2-Dose | Arm 5: NoV Vaccine Formulation A_1-Dose
Number analyzed (Participants) | 72 | 67 | 66 | 66 | 24
ratio
  Day 8: number analyzed (Participants) | 72 | 65 | 66 | 65 | 23
  Day 8 | 1.0 [0.9 to 1.1] | 10.1 [6.6 to 15.6] | 1.0 [0.9 to 1.0] | 14.1 [9.2 to 21.6] | 1.0 [0.9 to 1.0]
  Day 29: number analyzed (Participants) | 72 | 66 | 66 | 66 | 24
  Day 29 | 1.0 [1.0 to 1.0] | 13.0 [9.1 to 18.6] | 1.0 [1.0 to 1.1] | 12.0 [8.5 to 16.8] | 1.0 [0.9 to 1.1]
  Day 36: number analyzed (Participants) | 72 | 66 | 64 | 66 | 23
  Day 36 | 7.3 [4.9 to 10.9] | 12.6 [9.1 to 17.4] | 10.6 [7.0 to 15.9] | 14.2 [10.7 to 18.8] | 7.5 [3.9 to 14.6]
  Day 57: number analyzed (Participants) | 71 | 65 | 62 | 66 | 24
  Day 57 | 6.6 [4.8 to 9.1] | 12.1 [9.1 to 16.2] | 10.0 [7.1 to 14.0] | 13.3 [10.3 to 17.1] | 5.3 [3.0 to 9.6]
  Day 211: number analyzed (Participants) | 71 | 66 | 64 | 66 | 23
  Day 211 | 3.2 [2.6 to 4.0] | 5.5 [4.2 to 7.3] | 4.8 [3.7 to 6.3] | 5.3 [4.1 to 6.8] | 2.4 [1.4 to 4.0]
  Day 393: number analyzed (Participants) | 70 | 64 | 63 | 65 | 23
  Day 393 | 2.4 [1.9 to 3.0] | 3.9 [3.0 to 5.2] | 3.2 [2.5 to 4.1] | 3.5 [2.7 to 4.6] | 1.8 [1.1 to 2.9]

17. Secondary Outcome: GMFR of Anti-norovirus GII.4 VLP Antibody Titers (HBGA)
Description: GMFR of anti-norovirus GII.4 VLP antibody titers measured by HBGA blocking assay are reported. The fold rise was calculated as the ratio of the post-vaccination titer level to the pre-vaccination titer level.
Time Frame: Days 8, 29, 36, 57, 211 and 393
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Arm 1: NoV Vaccine Formulation A_1-Dose | Arm 2: NoV Vaccine Formulation A_2-Dose | Arm 3: NoV Vaccine Formulation B_1-Dose | Arm 4: NoV Vaccine Formulation B_2-Dose | Arm 5: NoV Vaccine Formulation A_1-Dose
Number analyzed (Participants) | 72 | 67 | 66 | 66 | 24
ratio
  Day 8: number analyzed (Participants) | 72 | 66 | 66 | 65 | 23
  Day 8 | 0.9 [0.8 to 1.0] | 6.9 [4.5 to 10.5] | 0.9 [0.8 to 1.1] | 11.6 [7.7 to 17.5] | 0.9 [0.8 to 1.0]
  Day 29 | 0.9 [0.8 to 1.0] | 7.9 [5.6 to 11.0] | 0.8 [0.7 to 1.0] | 10.2 [7.2 to 14.5] | 0.9 [0.8 to 1.0]
  Day 36: number analyzed (Participants) | 72 | 67 | 64 | 66 | 23
  Day 36 | 8.4 [5.4 to 13.0] | 7.5 [5.5 to 10.4] | 7.3 [4.8 to 11.2] | 9.3 [6.6 to 13.0] | 15.1 [7.1 to 32.2]
  Day 57: number analyzed (Participants) | 71 | 66 | 62 | 66 | 24
  Day 57 | 8.1 [5.8 to 11.4] | 5.8 [4.3 to 7.8] | 8.4 [6.1 to 11.7] | 7.1 [5.3 to 9.6] | 9.4 [4.8 to 18.4]
  Day 211: number analyzed (Participants) | 71 | 66 | 64 | 66 | 23
  Day 211 | 3.4 [2.6 to 4.5] | 3.0 [2.2 to 4.1] | 3.4 [2.5 to 4.5] | 3.7 [2.8 to 4.8] | 3.8 [2.2 to 6.5]
  Day 393: number analyzed (Participants) | 70 | 65 | 63 | 65 | 23
  Day 393 | 3.0 [2.3 to 3.8] | 2.6 [2.0 to 3.5] | 2.7 [2.1 to 3.5] | 3.2 [2.4 to 4.1] | 3.0 [1.7 to 5.4]

18. Secondary Outcome: Percentage of Participants With a 4-Fold Rise or Greater in Serum Anti-norovirus Antibody Titers for Both GI.1 VLP and GII.4 VLP as Measured by Total Immunoglobulin-Enzyme-linked Immunosorbent Assay (Pan-Ig ELISA)
Description: Percentage of participants with a 4-fold rise or greater in serum anti-norovirus antibody titers for both GI.1 VLP and GII.4 VLP measured by Pan-Ig ELISA are reported.
Time Frame: Days 8, 29, 36, 57, 211 and 393
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1: NoV Vaccine Formulation A_1-Dose | Arm 2: NoV Vaccine Formulation A_2-Dose | Arm 3: NoV Vaccine Formulation B_1-Dose | Arm 4: NoV Vaccine Formulation B_2-Dose | Arm 5: NoV Vaccine Formulation A_1-Dose
Number analyzed (Participants) | 72 | 67 | 66 | 66 | 24
percentage of participants
  Day 8: number analyzed (Participants) | 72 | 66 | 66 | 65 | 23
  Day 8 | 0.0 [0.0 to 5.0] | 31.8 [20.9 to 44.4] | 0.0 [0.0 to 5.4] | 52.3 [39.5 to 64.9] | 0.0 [0.0 to 14.8]
  Day 29 | 1.4 [0.0 to 7.5] | 47.8 [35.4 to 60.3] | 0.0 [0.0 to 5.4] | 62.1 [49.3 to 73.8] | 0.0 [0.0 to 14.2]
  Day 36: number analyzed (Participants) | 72 | 67 | 64 | 66 | 23
  Day 36 | 37.5 [26.4 to 49.7] | 49.3 [36.8 to 61.8] | 39.1 [27.1 to 52.1] | 63.6 [50.9 to 75.1] | 69.6 [47.1 to 86.8]
  Day 57: number analyzed (Participants) | 71 | 66 | 62 | 66 | 24
  Day 57 | 52.1 [39.9 to 64.1] | 43.9 [31.7 to 56.7] | 58.1 [44.8 to 70.5] | 62.1 [49.3 to 73.8] | 62.5 [40.6 to 81.2]
  Day 211: number analyzed (Participants) | 71 | 66 | 64 | 66 | 23
  Day 211 | 40.8 [29.3 to 53.2] | 37.9 [26.2 to 50.7] | 40.6 [28.5 to 53.6] | 42.4 [30.3 to 55.2] | 47.8 [26.8 to 69.4]
  Day 393: number analyzed (Participants) | 70 | 65 | 63 | 65 | 23
  Day 393 | 24.3 [14.8 to 36.0] | 15.4 [7.6 to 26.5] | 25.4 [15.3 to 37.9] | 23.1 [13.5 to 35.2] | 30.4 [13.2 to 52.9]

19. Secondary Outcome: Percentage of Participants With a 4-Fold Rise or Greater in Serum Anti-norovirus GI.1 VLP Antibody Titers (Pan-Ig ELISA)
Description: Percentage of participants with a 4-Fold rise or greater in serum anti-norovirus GI.1 VLP antibody titers measured by Pan-Ig ELISA are reported.
Time Frame: Days 8, 29, 36, 57, 211 and 393
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1: NoV Vaccine Formulation A_1-Dose | Arm 2: NoV Vaccine Formulation A_2-Dose | Arm 3: NoV Vaccine Formulation B_1-Dose | Arm 4: NoV Vaccine Formulation B_2-Dose | Arm 5: NoV Vaccine Formulation A_1-Dose
Number analyzed (Participants) | 72 | 67 | 66 | 66 | 24
percentage of participants
  Day 8: number analyzed (Participants) | 72 | 66 | 66 | 65 | 23
  Day 8 | 0.0 [0.0 to 5.0] | 56.1 [43.3 to 68.3] | 0.0 [0.0 to 5.4] | 69.2 [56.6 to 80.1] | 0.0 [0.0 to 14.8]
  Day 29 | 1.4 [0.0 to 7.5] | 67.2 [54.6 to 78.2] | 0.0 [0.0 to 5.4] | 80.3 [68.7 to 89.1] | 8.3 [1.0 to 27.0]
  Day 36: number analyzed (Participants) | 72 | 67 | 64 | 66 | 23
  Day 36 | 59.7 [47.5 to 71.1] | 67.2 [54.6 to 78.2] | 68.8 [55.9 to 79.8] | 83.3 [72.1 to 91.4] | 91.3 [72.0 to 98.9]
  Day 57: number analyzed (Participants) | 71 | 66 | 62 | 66 | 24
  Day 57 | 73.2 [61.4 to 83.1] | 65.2 [52.4 to 76.5] | 83.9 [72.3 to 92.0] | 84.8 [73.9 to 92.5] | 87.5 [67.6 to 97.3]
  Day 211: number analyzed (Participants) | 71 | 66 | 64 | 66 | 23
  Day 211 | 62.0 [49.7 to 73.2] | 63.6 [50.9 to 75.1] | 70.3 [57.6 to 81.1] | 72.7 [60.4 to 83.0] | 73.9 [51.6 to 89.8]
  Day 393: number analyzed (Participants) | 70 | 65 | 63 | 65 | 23
  Day 393 | 48.6 [36.4 to 60.8] | 41.5 [29.4 to 54.4] | 52.4 [39.4 to 65.1] | 60.0 [47.1 to 72.0] | 60.9 [38.5 to 80.3]

20. Secondary Outcome: Percentage of Participants With a 4-Fold Rise or Greater in Serum Anti-norovirus GII.4 VLP Antibody Titers (Pan-Ig ELISA)
Description: Percentage of participants with a 4-fold rise or greater in serum anti-norovirus GII.4 VLP antibody titers measured by Pan-Ig ELISA are reported.
Time Frame: Days 8, 29, 36, 57, 211 and 393
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1: NoV Vaccine Formulation A_1-Dose | Arm 2: NoV Vaccine Formulation A_2-Dose | Arm 3: NoV Vaccine Formulation B_1-Dose | Arm 4: NoV Vaccine Formulation B_2-Dose | Arm 5: NoV Vaccine Formulation A_1-Dose
Number analyzed (Participants) | 72 | 67 | 66 | 66 | 24
percentage of participants
  Day 8: number analyzed (Participants) | 72 | 66 | 66 | 65 | 23
  Day 8 | 0.0 [0.0 to 14.2] | 50.0 [29.1 to 70.9] | 0.0 [0.0 to 14.8] | 62.5 [40.6 to 81.2] | 0.0 [0.0 to 14.8]
  Day 29 | 0.0 [0.0 to 14.2] | 70.8 [48.9 to 87.4] | 0.0 [0.0 to 14.8] | 70.8 [48.9 to 87.4] | 0.0 [0.0 to 14.2]
  Day 36: number analyzed (Participants) | 72 | 67 | 64 | 66 | 23
  Day 36 | 52.8 [40.7 to 64.7] | 68.7 [56.2 to 79.4] | 48.4 [35.8 to 61.3] | 71.2 [58.7 to 81.7] | 73.9 [51.6 to 89.8]
  Day 57: number analyzed (Participants) | 71 | 66 | 62 | 66 | 24
  Day 57 | 70.4 [58.4 to 80.7] | 63.6 [50.9 to 75.1] | 67.7 [54.7 to 79.1] | 68.2 [55.6 to 79.1] | 66.7 [44.7 to 84.4]
  Day 211: number analyzed (Participants) | 71 | 66 | 64 | 66 | 23
  Day 211 | 60.6 [48.3 to 72.0] | 53.0 [40.3 to 65.4] | 50.0 [37.2 to 62.8] | 53.0 [40.3 to 65.4] | 52.2 [30.6 to 73.2]
  Day 393: number analyzed (Participants) | 70 | 65 | 63 | 65 | 23
  Day 393 | 34.3 [23.3 to 46.6] | 32.3 [21.2 to 45.1] | 34.9 [23.3 to 48.0] | 36.9 [25.3 to 49.8] | 34.8 [16.4 to 57.3]

21. Secondary Outcome: GMT of Anti-norovirus GI.1 VLP Antibody Titers (Pan-Ig ELISA)
Description: GMT of anti-norovirus GI.1 VLP antibody titers measured by Pan-Ig ELISA are reported.
Time Frame: Baseline (Day 1), Days 8, 29, 36, 57, 211 and 393
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Arm 1: NoV Vaccine Formulation A_1-Dose | Arm 2: NoV Vaccine Formulation A_2-Dose | Arm 3: NoV Vaccine Formulation B_1-Dose | Arm 4: NoV Vaccine Formulation B_2-Dose | Arm 5: NoV Vaccine Formulation A_1-Dose
Number analyzed (Participants) | 72 | 67 | 66 | 66 | 24
titer
  Baseline (Day 1) | 661.8 [508.5 to 861.2] | 906.1 [622.4 to 1319.3] | 838.5 [605.8 to 1160.4] | 619.7 [459.7 to 835.2] | 460.3 [204.8 to 1034.6]
  Day 8: number analyzed (Participants) | 72 | 66 | 66 | 65 | 23
  Day 8 | 678.0 [519.7 to 884.5] | 4534.9 [3303.2 to 6225.8] | 829.4 [603.0 to 1140.8] | 6382.8 [4698.1 to 8671.7] | 455.2 [192.4 to 1076.7]
  Day 29 | 668.2 [520.4 to 857.9] | 7701.1 [6141.9 to 9656.0] | 791.9 [585.7 to 1070.9] | 8951.5 [7127.3 to 11242.6] | 574.0 [273.1 to 1206.2]
  Day 36: number analyzed (Participants) | 72 | 67 | 64 | 66 | 23
  Day 36 | 4158.6 [3095.1 to 5587.6] | 7663.6 [6165.5 to 9525.6] | 6411.8 [4795.4 to 8573.1] | 9161.1 [7501.2 to 11188.4] | 7603.5 [4590.2 to 12595.1]
  Day 57: number analyzed (Participants) | 71 | 66 | 62 | 66 | 24
  Day 57 | 6183.5 [4929.9 to 7755.8] | 7235.1 [5945.9 to 8804.0] | 8838.3 [6928.3 to 11275.0] | 8182.2 [6751.1 to 9916.8] | 8165.5 [5659.8 to 11780.6]
  Day 211: number analyzed (Participants) | 71 | 66 | 64 | 66 | 23
  Day 211 | 3945.2 [3233.5 to 4813.6] | 5161.2 [4206.5 to 6332.6] | 5406.6 [4433.7 to 6593.0] | 4882.3 [4069.9 to 5856.9] | 3523.2 [2277.6 to 5449.9]
  Day 393: number analyzed (Participants) | 70 | 65 | 63 | 65 | 23
  Day 393 | 2903.4 [2307.1 to 3653.9] | 3672.1 [2835.7 to 4755.2] | 3862.9 [3060.2 to 4876.3] | 3370.0 [2799.0 to 4057.5] | 2252.6 [1365.3 to 3716.5]

22. Secondary Outcome: GMT of Anti-norovirus GII.4 VLP Antibody Titers (Pan-Ig ELISA)
Description: GMT of anti-norovirus GII.4 VLP antibody titers measured by Pan-Ig ELISA are reported.
Time Frame: Baseline (Day 1), Days 8, 29, 36, 57, 211 and 393
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Arm 1: NoV Vaccine Formulation A_1-Dose | Arm 2: NoV Vaccine Formulation A_2-Dose | Arm 3: NoV Vaccine Formulation B_1-Dose | Arm 4: NoV Vaccine Formulation B_2-Dose | Arm 5: NoV Vaccine Formulation A_1-Dose
Number analyzed (Participants) | 72 | 67 | 66 | 66 | 24
titer
  Baseline (Day 1) | 761.9 [547.9 to 1059.7] | 1054.9 [707.8 to 1572.4] | 1066.3 [719.7 to 1580.0] | 897.4 [612.3 to 1315.3] | 1023.2 [543.8 to 1925.3]
  Day 8: number analyzed (Participants) | 72 | 66 | 66 | 65 | 23
  Day 8 | 766.6 [553.1 to 1062.6] | 4725.5 [3479.7 to 6417.3] | 1078.9 [726.6 to 1602.0] | 5691.9 [4107.9 to 7886.7] | 1054.6 [550.6 to 2020.2]
  Day 29 | 766.8 [553.7 to 1062.0] | 8105.1 [6053.8 to 10851.6] | 1017.7 [690.1 to 1500.8] | 8314.1 [6388.3 to 10820.3] | 1022.4 [574.4 to 1819.7]
  Day 36: number analyzed (Participants) | 72 | 67 | 64 | 66 | 23
  Day 36 | 4587.6 [3402.2 to 6186.0] | 7911.9 [6059.9 to 10329.8] | 5411.9 [3777.0 to 7754.5] | 8025.5 [6339.1 to 10160.5] | 10084.9 [7037.2 to 14452.5]
  Day 57: number analyzed (Participants) | 71 | 66 | 62 | 66 | 24
  Day 57 | 6564.1 [5151.3 to 8364.5] | 7489.2 [5788.1 to 9690.4] | 7877.2 [5878.8 to 10554.9] | 7028.4 [5611.6 to 8803.0] | 9507.3 [7110.9 to 12711.2]
  Day 211: number analyzed (Participants) | 71 | 66 | 64 | 66 | 23
  Day 211 | 3702.0 [2913.0 to 4704.7] | 4915.8 [3676.9 to 6572.2] | 4657.8 [3510.6 to 6179.8] | 4456.2 [3493.1 to 5684.9] | 4531.5 [3194.5 to 6428.0]
  Day 393: number analyzed (Participants) | 70 | 65 | 63 | 65 | 23
  Day 393 | 2216.7 [1708.9 to 2875.3] | 3151.5 [2319.8 to 4281.5] | 2807.4 [2081.9 to 3785.8] | 2853.9 [2225.5 to 3659.7] | 2969.5 [1818.4 to 4849.5]

23. Secondary Outcome: GMFR of Anti-norovirus GI.1 VLP Antibody Titers (Pan-Ig ELISA)
Description: GMFR of anti-norovirus GI.1 VLP antibody titers measured by Pan-Ig ELISA are reported. The fold rise was calculated as the ratio of the post-vaccination titer level to the pre-vaccination titer level.
Time Frame: Days 8, 29, 36, 57, 211 and 393
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Arm 1: NoV Vaccine Formulation A_1-Dose | Arm 2: NoV Vaccine Formulation A_2-Dose | Arm 3: NoV Vaccine Formulation B_1-Dose | Arm 4: NoV Vaccine Formulation B_2-Dose | Arm 5: NoV Vaccine Formulation A_1-Dose
Number analyzed (Participants) | 72 | 67 | 66 | 66 | 24
ratio
  Day 8: number analyzed (Participants) | 72 | 66 | 66 | 65 | 23
  Day 8 | 1.0 [1.0 to 1.1] | 5.1 [3.7 to 7.2] | 1.0 [0.9 to 1.0] | 10.3 [7.2 to 14.7] | 1.0 [0.9 to 1.1]
  Day 29 | 1.0 [0.9 to 1.1] | 8.5 [6.2 to 11.7] | 0.9 [0.9 to 1.0] | 14.4 [10.7 to 19.5] | 1.2 [0.9 to 1.8]
  Day 36: number analyzed (Participants) | 72 | 67 | 64 | 66 | 23
  Day 36 | 6.3 [4.5 to 8.8] | 8.5 [6.1 to 11.7] | 7.6 [5.5 to 10.6] | 14.8 [10.9 to 20.0] | 17.3 [8.4 to 35.9]
  Day 57: number analyzed (Participants) | 71 | 66 | 62 | 66 | 24
  Day 57 | 9.0 [6.8 to 11.9] | 7.9 [5.8 to 10.8] | 11.4 [8.3 to 15.6] | 13.2 [9.9 to 17.7] | 17.7 [8.8 to 35.8]
  Day 211: number analyzed (Participants) | 71 | 66 | 64 | 66 | 23
  Day 211 | 6.0 [4.8 to 7.5] | 5.8 [4.3 to 7.7] | 6.4 [4.9 to 8.5] | 7.9 [6.2 to 10.0] | 8.0 [4.1 to 15.4]
  Day 393: number analyzed (Participants) | 70 | 65 | 63 | 65 | 23
  Day 393 | 4.4 [3.6 to 5.5] | 4.0 [3.1 to 5.3] | 4.6 [3.6 to 5.9] | 5.2 [4.2 to 6.5] | 5.1 [2.6 to 10.1]

24. Secondary Outcome: GMFR of Anti-norovirus GII.4 VLP Antibody Titers (Pan-Ig ELISA)
Description: GMFR of anti-norovirus GII.4 VLP antibody titers measured by Pan-Ig ELISA are reported. The fold rise was calculated as the ratio of the post-vaccination titer level to the pre-vaccination titer level.
Time Frame: Days 8, 29, 36, 57, 211 and 393
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Arm 1: NoV Vaccine Formulation A_1-Dose | Arm 2: NoV Vaccine Formulation A_2-Dose | Arm 3: NoV Vaccine Formulation B_1-Dose | Arm 4: NoV Vaccine Formulation B_2-Dose | Arm 5: NoV Vaccine Formulation A_1-Dose
Number analyzed (Participants) | 72 | 67 | 66 | 66 | 24
ratio
  Day 8: number analyzed (Participants) | 72 | 66 | 66 | 65 | 23
  Day 8 | 1.0 [1.0 to 1.1] | 4.5 [3.2 to 6.2] | 1.0 [1.0 to 1.1] | 6.3 [4.5 to 9.0] | 1.0 [0.9 to 1.0]
  Day 29 | 1.0 [0.9 to 1.1] | 7.7 [5.7 to 10.4] | 1.0 [0.9 to 1.0] | 9.3 [6.7 to 12.8] | 1.0 [0.9 to 1.1]
  Day 36: number analyzed (Participants) | 72 | 67 | 64 | 66 | 23
  Day 36 | 6.0 [4.3 to 8.4] | 7.5 [5.6 to 10.0] | 5.0 [3.6 to 6.9] | 8.9 [6.4 to 12.4] | 9.6 [5.1 to 18.1]
  Day 57: number analyzed (Participants) | 71 | 66 | 62 | 66 | 24
  Day 57 | 8.7 [6.4 to 11.7] | 6.9 [5.2 to 9.2] | 8.3 [6.2 to 11.0] | 7.8 [5.8 to 10.6] | 9.3 [5.1 to 16.8]
  Day 211: number analyzed (Participants) | 71 | 66 | 64 | 66 | 23
  Day 211 | 4.9 [3.8 to 6.3] | 4.6 [3.6 to 5.9] | 4.5 [3.5 to 5.7] | 5.0 [3.8 to 6.4] | 4.7 [3.0 to 7.5]
  Day 393: number analyzed (Participants) | 70 | 65 | 63 | 65 | 23
  Day 393 | 3.1 [2.4 to 3.8] | 3.1 [2.4 to 3.9] | 2.6 [2.1 to 3.3] | 3.0 [2.4 to 3.8] | 3.1 [1.9 to 5.0]

25. Secondary Outcome: Percentage of Participants With At Least One Adverse Event of Special Interest (AESI)
Description: AESIs are AEs that are not solicited local or systemic AEs, they are predefined AEs that required close monitoring and prompt reporting to the sponsor. AESI included protocol specified Cardiac Disorders, Gastrointestinal Disorders, Immune System Disorders, Infections and Infestations, Musculoskeletal and Connective Tissue Diseases, Neuroinflammatory Disorders, Renal and Urinary Disorders, Skin Disorders, Thyroid Disorders, Vascular Disorders and Other Disorders.
Time Frame: From first vaccination up to Day 393
Population: SAF included all participants who received at least 1 dose of vaccine (NoV VLP vaccine or placebo).
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: NoV Vaccine Formulation A_1-Dose | Arm 2: NoV Vaccine Formulation A_2-Dose | Arm 3: NoV Vaccine Formulation B_1-Dose | Arm 4: NoV Vaccine Formulation B_2-Dose | Arm 5: NoV Vaccine Formulation A_1-Dose
Number analyzed (Participants) | 76 | 74 | 72 | 72 | 25
percentage of participants | 1.3 | 2.7 | 2.8 | 0.0 | 0.0

26. Secondary Outcome: Percentage of Participants With At Least One Adverse Event (AE) Leading to Participant's Withdrawal From the Study
Description: Withdrawal due to an AE will occur if the participant experiences an AE that requires early termination of treatment, because continued participation imposes an unacceptable risk to the participant's health or the participant is unwilling to continue because of the AE.
Time Frame: From first vaccination up to Day 393
Population: SAF included all participants who received at least 1 dose of vaccine (NoV VLP vaccine or placebo).
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: NoV Vaccine Formulation A_1-Dose | Arm 2: NoV Vaccine Formulation A_2-Dose | Arm 3: NoV Vaccine Formulation B_1-Dose | Arm 4: NoV Vaccine Formulation B_2-Dose | Arm 5: NoV Vaccine Formulation A_1-Dose
Number analyzed (Participants) | 76 | 74 | 72 | 72 | 25
percentage of participants | 1.3 | 1.4 | 0.0 | 1.4 | 0.0

ADVERSE EVENTS:
Time Frame: All-Cause Mortality and Serious adverse events: From first vaccination (Day 1) through end of study (Day 393); Other adverse events: From any vaccination (Day 1 and Day 29) up to 28 days post vaccination.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. SAF included all participants who received at least 1 dose of vaccine (NoV VLP vaccine or placebo).
Arm/Group | Arm 1: NoV Vaccine Formulation A_1-Dose | Arm 2: NoV Vaccine Formulation A_2-Dose | Arm 3: NoV Vaccine Formulation B_1-Dose | Arm 4: NoV Vaccine Formulation B_2-Dose | Arm 5: NoV Vaccine Formulation A_1-Dose
All-Cause Mortality (participants affected / at risk) | 1/76 | 1/74 | 0/72 | 1/72 | 0/25
Serious Adverse Events (participants affected / at risk) | 7/76 | 9/74 | 17/72 | 9/72 | 0/25
Other Adverse Events (participants affected / at risk) | 28/76 | 25/74 | 23/72 | 21/72 | 7/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: NoV Vaccine Formulation A_1-Dose (N=76) | Arm 2: NoV Vaccine Formulation A_2-Dose (N=74) | Arm 3: NoV Vaccine Formulation B_1-Dose (N=72) | Arm 4: NoV Vaccine Formulation B_2-Dose (N=72) | Arm 5: NoV Vaccine Formulation A_1-Dose (N=25)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 2 | 1 | 0
Aortic valve stenosis (Cardiac disorders) | 1 | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Stress cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 1 | 0 | 0
Complication associated with device (General disorders) | 0 | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Splenic abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Streptococcal endocarditis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 0 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 — One treatment-emergent death occurred during treatment with NoV vaccine (formulation B)-2 dose regimen and is not related. Same participant had metabolic encephalopathy and ruptured cerebral aneurysm.
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 — One treatment-emergent death occurred during treatment with NoV vaccine (formulation B)-2 dose regimen and is not related. Same participant had haemorrhagic stroke and ruptured cerebral aneurysm.
Ruptured cerebral aneurysm (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 — One treatment-emergent death occurred during treatment with NoV vaccine (formulation B)-2 dose regimen and is not related. Same participant had haemorrhagic stroke and metabolic encephalopathy.
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 — One treatment-emergent death occurred during treatment with NoV vaccine (formulation A)-2 dose regimen and is not related.
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 — One treatment-emergent death occurred during treatment with NoV vaccine (formulation A)-1 dose regimen and is not related.
Bladder outlet obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: NoV Vaccine Formulation A_1-Dose (N=76) | Arm 2: NoV Vaccine Formulation A_2-Dose (N=74) | Arm 3: NoV Vaccine Formulation B_1-Dose (N=72) | Arm 4: NoV Vaccine Formulation B_2-Dose (N=72) | Arm 5: NoV Vaccine Formulation A_1-Dose (N=25)
Upper respiratory tract infection (Infections and infestations) | 8 | 8 | 5 | 3 | 1
Viral upper respiratory tract infection (Infections and infestations) | 2 | 4 | 0 | 1 | 2
Bronchitis (Infections and infestations) | 0 | 1 | 2 | 2 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 2 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Injection site bruising (General disorders) | 4 | 1 | 4 | 2 | 0
Fatigue (General disorders) | 3 | 3 | 1 | 3 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 3 | 2 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 2 | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 2 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 1
Exposure to communicable disease (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 2 | 3 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 3 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 2 | 1
Poor quality sleep (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0
Hypertension (Vascular disorders) | 2 | 0 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-02-02): https://cdn.clinicaltrials.gov/large-docs/90/NCT02661490/SAP_000.pdf
  • Study Protocol (2015-11-16): https://cdn.clinicaltrials.gov/large-docs/90/NCT02661490/Prot_001.pdf